CLINICAL TRIAL: NCT02075671
Title: Photodynamic Therapy for Papulopustular Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 031416
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Rosacea; Papulopustular Rosacea
Keywords: Rosacea; Photodynamic Therapy; Aminolevulinic Acid; Papulopustular Rosacea; Blue Light
MeSH Terms: conditions — Rosacea | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levulan and Blu-U Light (Experimental): Entire face treated with 20% Aminolevulinic Acid (Levulan) and Blu-U light
  Interventions: Drug: Aminolevulinic acid topical solution 20%; Device: Blu-U Light Therapy
- Vehicle and Blu-U Light (Sham Comparator): Entire face treated with vehicle substance only and Blu-U light
  Interventions: Device: Blu-U Light Therapy
- Vehicle Only (Placebo Comparator): Entire face treated with vehicle substance only
  Interventions: Other: Placebo vehicle only

INTERVENTIONS:
Drug: Aminolevulinic acid topical solution 20% — Intervention used in the experimental arm only
  Other Names: Levulan Kerastick
  Arms: Levulan and Blu-U Light
Device: Blu-U Light Therapy — Intervention used in experimental and sham arms
  Arms: Levulan and Blu-U Light; Vehicle and Blu-U Light
Other: Placebo vehicle only — Intervention only includes the placebo vehicle solution
  Arms: Vehicle Only

SUMMARY:
Rosacea is a chronic inflammatory disorder that is characterized by severe flushing (transient erythema), non-transient erythema, papules, pustules, and telangiectasia. Topical therapy is not always effective in treating symptoms of rosacea. Furthermore, rapid recurrence is common following the use of systemic antibiotics, resulting in the chronic use of these medications to control the disease. Although the exact pathogenesis of rosacea is unknown, treatment for this condition has been investigated based on its similarity to acne and photodamaged skin. Case reports have shown promising results in rosacea patients treated with methyl aminolevulinate photodynamic therapy (MAL - PDT). Other than a case report which observed significant improvement of papules, pustules, erythema, and flushing following 5 - aminolevulinic acid photodynamic therapy (ALA-PDT) treatment of a patient with rosacea, the role of ALA-PDT in the treatment of rosacea has not been reported.

We have designed a pilot study investigating the efficacy of ALA-PDT in treating papulopustular rosacea. The objectives of the study are as follows:

Primary objective:

1. To evaluate improvement of the inflammatory lesions (papules, pustules, nodules), erythema, and telangiectasia of rosacea as assessed by the Investigator's Global Assessment (IGA).
2. To evaluate improvement of the inflammatory lesions (papules, pustules, nodules) of rosacea as assessed by the Inflammatory Lesion Investigator's Global Assessment (ILIGA).

   Secondary objectives:
3. To evaluate improvement of rosacea associated erythema as assessed by the Clinical Erythema Assessment (CEA) scale.
4. To evaluate improvement of the inflammatory lesions (papules, pustules, nodules) of rosacea as measured by a difference in inflammatory lesion count.
5. To evaluate improvement of rosacea as assessed by the Patient Overall Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-79 years
2. Clinical diagnosis of papulopustular rosacea based on physician evaluation. Only patients with 3-50 papules and/or pustules, and a CEA total score ≥ 5, (See Section 4.1.3) will be enrolled.
3. History of failing at least one conventional treatment for rosacea (metronidazole, sodium sulfacetamide, tetracycline, azelaic acid) or not interested in continuous treatment with these agents.

Exclusion Criteria:

1. < 18 or > 79 years of age
2. Allergy to 5 - aminolevulinic acid (ALA) or any component of the vehicle
3. Use of topical acne or rosacea treatments (on the face) within 2 weeks prior to Visit 1
4. Use of systemic antibiotics within 1 month prior to Visit 1
5. Use of topical retinoids (on the face) within 1 month prior to Visit 1
6. Use of systemic retinoids, including isotretinoin, within 6 months prior to Visit 1.
7. Use of laser or light based rosacea treatments (on the face) within 1 month prior to Visit 1
8. Cosmetic procedures (e.g., superficial chemical peels, exfoliation or microdermabrasion of the face) within 2 months prior to Visit 1
9. Use of topical corticosteroids (on the face) 1 month prior to Visit 1
10. Use of systemic corticosteroids 3 months prior to Visit 1
11. Known or suspected history of drug or alcohol abuse within the past 6 months as determined by the medical record or patient interview
12. History of adverse reaction to light exposure
13. History of disorder of porphyrin metabolism
14. Scarring or infection in the area being treated
15. Extensive facial hair that would either impair blue light exposure or interfere with lesion evaluation
16. Inability to make study visits or anticipated poor compliance
17. Pregnant females or nursing mothers. Eligible women of reproductive age will be required to have a negative urine pregnancy test at screening. They will also be required to be on at least one reliable form of effective birth control [examples: barrier method (condoms, diaphragm), oral, injectable, implant birth control or abstinence] during the course of this study and 30 days following the last treatment period.
18. Life threatening illness that would interfere with the patient's ability to complete the study
19. Participation in another clinical experimental therapeutic study within 30 days of screening visit
20. Any history or evidence of severe illness or any other condition that would make the patient, in the opinion of the investigator, unsuitable for the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Ehrlich, MD, MHS, Principal Investigator — George Washington University Department of Dermatology; Kamaria Nelson, MD, Study Director — George Washington University Department of Dermatology
Locations (1):
- Medical Faculty Associates - George Washington University, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levulan and Blu-U Light | Vehicle and Blu-U Light | Vehicle Only
Started | 10 | 10 | 10
Completed | 8 | 10 | 6
Not Completed | 2 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levulan and Blu-U Light | Vehicle and Blu-U Light | Vehicle Only | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 9 | 28
  >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 24
  Male | 1 | 3 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 9 | 9 | 10 | 28
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick classification is a method of skin phototyping based on a person's tendency to sunburn and ability to tan.
  I: Always burn, never tan II: Usually burn, tan less than average (with difficulty) III: Sometimes mild burn, tan about average IV: Rarely burn, tan more than average (with ease) V: Brown skin VI: Black skin
  Participants
    I | 2 | 6 | 1 | 9
    II | 5 | 4 | 9 | 18
    III | 2 | 0 | 0 | 2
    IV | 0 | 0 | 0 | 0
    V | 1 | 0 | 0 | 1
    VI | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Improvement of the Inflammatory Lesions (Papules, Pustules, Nodules), Erythema, and Telangiectasia of Rosacea as Assessed by the Investigator's Global Assessment (IGA)
Description: The Investigator's global assessment (IGA) of rosacea is a subjective 7-point, static scoring system. Scores range from 0 to 6: 0 (clear), 1 (minimal), 2 (mild), 3 (mild to moderate), 4 (moderate), 5 (moderate to severe), 6 (severe).
Time Frame: 17 weeks
Population: Group A = Levulan and Blu-U Light; Group B = Vehicle and Blu-U Light; Group C = Vehicle Only. Of the 30 randomized patients, 24 (80%) completed the entire study. 8 (80%) patients completed from Group A, 10 (100%) from Group B, and 6 (60%) from Group C.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levulan and Blu-U Light | Vehicle and Blu-U Light | Vehicle Only
Number analyzed (Participants) | 8 | 10 | 6
score on a scale | 2.8 (0.5) | 1.5 (1.6) | 1.5 (0.8)

2. Primary Outcome: Improvement of the Inflammatory Lesions (Papules, Pustules, Nodules) of Rosacea as Assessed by the Inflammatory Lesion Investigator's Global Assessment (ILIGA)
Description: The Inflammatory Lesion Investigator's Global Assessment (ILIGA) is a subjective 5-point measure of the overall disease severity. Scores range from 0 to 4: 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate), 4 (severe).
Time Frame: 17 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levulan and Blu-U Light | Vehicle and Blu-U Light | Vehicle Only
Number analyzed (Participants) | 8 | 10 | 6
score on a scale | 1.3 (0.9) | 0.8 (1.2) | 1.0 (0.9)

3. Secondary Outcome: Evaluate Improvement of Rosacea Associated Erythema as Assessed by the Clinical Erythema Assessment (CEA) Scale
Description: The Clinical Erythema Assessment (CEA) scale is an assessment of erythema. It has a score range from 0 to 4: 0 (none), 1 (mild), 2 (moderate), 3 (significant), 4 (severe). The total score is based on the evaluation of all areas of the face (forehead, chin, right cheek, left cheek, and nose). Each of these areas were scored from 0-4, giving a maximum total score of 20.
Time Frame: 17 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levulan and Blu-U Light | Vehicle and Blu-U Light | Vehicle Only
Number analyzed (Participants) | 8 | 10 | 6
score on a scale | 6.0 (2.1) | 4.5 (3.6) | 1.2 (3.9)

4. Secondary Outcome: Evaluate Improvement of the Inflammatory Lesions (Papules, Pustules, Nodules) of Rosacea as Measured by a Difference in Inflammatory Lesion Count (ILC)
Description: The Inflammatory Lesion Count (ILC) is calculated by the number of inflammatory lesions (papules, pustules, nodules) as recorded by the investigator.
Time Frame: 17 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Inflammatory Lesion Count
Arm/Group | Levulan and Blu-U Light | Vehicle and Blu-U Light | Vehicle Only
Number analyzed (Participants) | 8 | 10 | 6
Inflammatory Lesion Count | 10.8 (2.9) | 3.4 (7.0) | 6.2 (5.0)

5. Secondary Outcome: Evaluate Improvement of Rosacea as Assessed by the Patient Overall Assessment (POA) Scale
Description: For the Patient Overall Assessments (POA) scale, patients assessed the overall improvement of their rosacea using a 4-point scale, where 1 = excellent improvement, 2 = good/moderate improvement, 3 = no change, 4 = worsening.
Time Frame: 17 weeks
Population: Group A = Levulan and Blu-U Light; Group B = Vehicle and Blu-U Light; Group C = Vehicle Only. 8 (80%) patients completed from Group A, 10 (100%) from Group B, and 6 (60%) from Group C. One participant in Group B did not complete the POA scale at the last follow-up visit; therefore only 9 participants are included in the analysis for Group B.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levulan and Blu-U Light | Vehicle and Blu-U Light | Vehicle Only
Number analyzed (Participants) | 8 | 9 | 6
score on a scale | 0.9 (1.0) | 0.6 (0.9) | 0.3 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for each patient from the baseline visit to up to 2 months following the final treatment, which averages from 17 to 19 weeks per patient.
Arm/Group | Levulan and Blu-U Light | Vehicle and Blu-U Light | Vehicle Only
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 0/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levulan and Blu-U Light (N=10) | Vehicle and Blu-U Light (N=10) | Vehicle Only (N=10)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
Post-Treatment Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT02075671/Prot_SAP_000.pdf